CLINICAL TRIAL: NCT01725373
Title: Prospective Registry in Patients With Unprotected Left Main Disease Treated by Percutaneous Coronary Intervention: The ALMA (Angioplasty of Left Main - lAriboisiere) Registry
Brief Title: Angioplasty of Left Main - lAriboisiere Registry
Acronym: ALMA
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Dr Jean-Guillaume DILLINGER, Principal investigator - Medical Doctor in the Departement of Cardiology, Hopital Lariboisière
Other Study IDs: LRB-06-012
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Artery Disease
Keywords: left main, stent,angioplasty
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Angioplasty of left main: Patients with:
  * stable or unstable angina and/or documented ischemia
  * de novo ≥50% stenosis in the left main stem referred for angioplasty

SUMMARY:
In patients with unprotected left main disease (ULMD), angioplasty is emerging as an alternative technique. The investigators aimed to determine the rate of major cardiovascular events in patients treated by angioplasty for ULMD in a "real world" registry.

DETAILED DESCRIPTION:
Current guidelines recommend coronary artery bypass graft surgery as the "gold standard" treatment in patients with unprotected left main disease. However, patients with ULMD and high surgical risk score or favourable anatomy are still referred for angioplasty. Recently, several studies and registries comparing surgery and percutaneous intervention with drug eluting stents report similar results regarding cardiovascular death and myocardial infarction in patients with multivessel coronary artery disease including unprotected left main disease.

The aim of the study is to evaluate major cardiovascular events in a "real world" registry.

ELIGIBILITY:
Inclusion Criteria:

* stable or unstable angina and/or documented ischemia
* 50% de novo ULMD referred for angioplasty

Exclusion Criteria:

* acute coronary syndrome with ST elevation,
* cardiogenic shock or out of hospital cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with stenosis of unprotected left main and schedulded angioplasty in the Department of Cardiology, Lariboisiere Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2007-01; Primary Completion 2012-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular events (MACCE) | One year
  Major cardiovascular events (MACCE)were measured after 1 year follow-up. MACCE included all-cause of death, stroke, myocardial infarction, and repeat revascularizations. Non-Q-wave myocardial infarction was defined using universal definition with troponin I. Stent thrombosis was defined according to the Academic Research Consortium definition as definite, probable, or possible and as early or late after the index procedure. Repeat revascularization was composed of any repeat percutaneous intervention or surgical bypass.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Henry, MD-PhD, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- Departement of Cardiology, Laribosiere Hospital, APHP, Paris, France